CLINICAL TRIAL: NCT03215251
Title: Experimental Study to Evaluate the Effectiveness of an Intervention Bundle on Thirst Intensity and Dry Mouth Among Patients of Selected Units
Brief Title: Effectiveness of an Intervention Bundle on Thirst Intensity and Dry Mouth Among Patients in ICUs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Shikha Gulia, Student, M.Sc Nursing, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 773
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Thirst; Dry Mouth
Keywords: Thirst, Dry Mouth, Intervention Bundle
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): Intervention bundle consisted of sterile cold wet oral swab wipes and sterile ice cold water sprays administered in two sessions of 15 minutes each. First session was given in 15 minutes, patients received cold wet oral swab wipes in oral cavity 2 to 3 times and mouth spray with 5 to 6 sprays. A maximum of 9 wipes and 18 sprays of sterile water. After administration of intervention bundle, Posttest 1 was taken after 15 minutes observation with the same tools. Then researcher waited for 15 minutes after post test1 and session two was administered in 15 minutes with a maximum of 9 wipes and 18 sprays of sterile water. Post test 2 was taken after 15 minutes of session two.
  Interventions: Other: Intervention bundle
- CONTROL GROUP (No Intervention): No Intervention administered. Thirst and Dry mouth scores were assessed only. Usual care was continued.

INTERVENTIONS:
Other: Intervention bundle — Assessment of the patient's mouth and lips determined, to check any stickiness or dryness in the mouth or around lips or split skin at the corners of the mouth or cracked lips. Intervention bundle consisted of sterile cold wet oral swab wipes and sterile ice cold water sprays administered for in two sessions of 15 minutes each. First session was given in 15 minutes, patients received cold wet oral swab wipes in oral cavity 2 to 3 times and mouth spray with 5 to 6 sprays. A maximum of 9 wipes and 18 sprays of sterile water. After administration of intervention bundle, Posttest 1 was taken after 15 minutes observation with the same tools. Then researcher waited for 15 minutes after post test1 and session two was administered in 15 minutes with a maximum of 9 wipes and 18 sprays of sterile water. Post test 2 was taken after 15 minutes of session two.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
The study evaluates the effectiveness of an Intervention Bundle on Thirst Intensity and Dry Mouth among Patients admitted in ICUs. Patients were randomized into two groups - Experimental and Control group. Experimental group received intervention Bundle whereas control group didn't receive any intervention. Usual care was continued in both the groups.

DETAILED DESCRIPTION:
The Convenience sampling technique was used to select Maharishi Markandeshwar institution of Medical Science and Researches Hospital, Mullana, Ambala. Intensive Care Units and a total of 60 patients in those units were also selected conveniently. The selected patients were randomly assigned to experimental and control group using lottery method. The total sample size for the study was 60 patients i.e. - 30 in experimental group and 30 in control group.

Experimental Group -patients were explained regarding administration of intervention bundle.Assessment of patients' mouth and lips was determined firstly. Intervention bundle consisted of sterile cold wet oral swab wipes and sterile ice cold water sprays administered for in two sessions of 15 minutes each. First session was given in 15 minutes, patients received cold wet oral swab wipes in oral cavity 2 to 3 times and mouth spray with 5 to 6 sprays. A maximum of 9 wipes and 18 sprays of sterile water. After administration of intervention bundle, Post test 1 was taken after 15 minutes observation with the same tools. Then researcher waited for 15 minutes after post test1 and session two was administered in 15 minutes with a maximum of 9 wipes and 18 sprays of sterile water. Post test 2 was taken after 15 minutes of session two.

Control group: control group was not given any intervention. Sample characteristics and clinical data (variables) were recorded in record sheet and thirst intensity and dry mouth scores were assessed only. After 30 minutes of pre test scores, post test 1 was taken and data were recorded. Then after, 30 minutes of post test 1, post test 2 was taken and data were recorded.

(Intervention to the control group was given after accomplishment of Post test for ethical consideration).

ELIGIBILITY:
Inclusion Criteria:

1. 18 or above 18 years of age.
2. Having thirst score ≥ 5 and dry mouth score ≥ 1
3. Willing to participate in the study.
4. Able to report verbally or non verbally about thirst intensity.
5. Admitted in ICCU,Respiratory ICU, Neurosurgical ICU and step Up ICU

Exclusion Criteria:

1. On mechanical ventilation.
2. Not able to follow the commands.
3. Having any oral surgery
4. Having open sores or desquamation of mouth and lips

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Thirst intensity Scale | 10 minutes
  To assess thirst intensity
  The scoring in the scale is given :
  1. not thirsty at all
  2. not very thirsty
  3. not thirsty
  4. neutral
  5. thirsty
  6. very thirsty
  7. very very thirsty
Dry Mouth assessment scale | 5 minutes
  to assess dry mouth

CONTACTS AND LOCATIONS:
Overall Officials: Mrs. Vinay Kumari, M.Sc Nursing, Study Director — M.M University, Mullana, Ambala, Haryana, India

REFERENCES:
- [Background] Puntillo K, Arai SR, Cooper BA, Stotts NA, Nelson JE. A randomized clinical trial of an intervention to relieve thirst and dry mouth in intensive care unit patients. Intensive Care Med. 2014 Sep;40(9):1295-302. doi: 10.1007/s00134-014-3339-z. Epub 2014 Jun 4. PMID 24894026
- [Background] Arai SR, Butzlaff A, Stotts NA, Puntillo KA. Quench the thirst: lessons from clinical thirst trials. Biol Res Nurs. 2014 Oct;16(4):456-66. doi: 10.1177/1099800413505900. Epub 2013 Oct 16. PMID 24136996
- [Background] Nelson JE, Meier DE, Oei EJ, Nierman DM, Senzel RS, Manfredi PL, Davis SM, Morrison RS. Self-reported symptom experience of critically ill cancer patients receiving intensive care. Crit Care Med. 2001 Feb;29(2):277-82. doi: 10.1097/00003246-200102000-00010. PMID 11246306
- [Result] Stotts NA, Arai SR, Cooper BA, Nelson JE, Puntillo KA. Predictors of thirst in intensive care unit patients. J Pain Symptom Manage. 2015 Mar;49(3):530-8. doi: 10.1016/j.jpainsymman.2014.07.001. Epub 2014 Aug 10. PMID 25116914